CLINICAL TRIAL: NCT01294839
Title: Right Ventricular Outflow Tract Septal Pacing for Cardiac Dysfunction Prevention Evaluation
Brief Title: Right Ventricular Outflow Tract Study
Acronym: RVOTCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-10-016-AP-LV
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Sinus-node Dysfunction
Keywords: sinus-node dysfunction; RVOTs pacing; RVA pacing
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RVOTs (Experimental): 555 Patients will be randomized to three groups(RVOTs, RVA, AAI) in 1:1:1, 185 patients in RVOTs arm, the RV lead of this group patients will be implanted in right ventricular outflow tract septum,the accumulated ventricular pacing percentage should be over 80% by adjusting AV delays.
  Interventions: Device: Right ventricular lead location
- AAI (Experimental): 555 Patients will be randomized to three groups(RVOTs, RVA, AAI) in 1:1:1, 185 patients in AAI arm, the RV lead of this group patients will be implanted in right ventricular apex.
  Interventions: Device: Right ventricular lead location
- RVA (Active Comparator): 555 Patients will be randomized to three groups(RVOTs, RVA, AAI) in 1:1:1, 185 patients in RVA arm, the RV lead of this group patients will be implanted in right ventricular apex, the accumulated ventricular pacing percentage should be over 80% by adjusting AV delays.
  Interventions: Device: Right ventricular lead location

INTERVENTIONS:
Device: Right ventricular lead location — RV leads in RVOTs group will be located in right ventricular outflow tract septum, RV leads in the other two group will be implanted in right ventricular apex, for the last RVOTs and RVA groups, the accumulated ventricular pacrouping percentage should be over 80% by adjusting AV delays.

SUMMARY:
This is a prospective, randomized, double blinded, multi-center, controlled study to evaluate the clinical impact at 18 months after DDD implantation of alternative pacing site (RVOTs and RVA) and the different conduction path (RVOTs and AV node) on cardiac dysfunction prevention.

DETAILED DESCRIPTION:
Ventricular pacing is unavoidable in many patients because of unreliable or absent AV conduction, or permanent AF. In recognition of this need, interest has focused on alternative site(s) ventricular pacing to maximize pumping function. These sites include the RV septum, His bundle, various LV sites, and combination of LV and RV (biventricular [BiV]). The RV outflow tract septum (RVOTs) seems to be the most promising site within the RV.

However, small enrollment and inconsistent experimental methods hinder the interpretation of these studies. Locations of alternative pacing sites were not clearly specified, were largely topographic, and lacked consistent anatomic designation. And what is more, there was no prospective, double-blind randomized, multi-center clinical trial which is design to test whether RVOTs pacing is superior to right ventricular apical pacing in preserving left ventricular systolic function and avoiding adverse left ventricular remodeling in patients with a normal left ventricular ejection fraction, ventricular synchrony and standard indications for pacing (sinus node dysfunction) in China. There was also no prospective, double-blind randomized, multi-center clinical trial which is design to test whether RVOTs pacing is not inferior to AAIR pacing in preserving left ventricular systolic function and avoiding adverse left ventricular remodeling in patients with a normal left ventricular ejection fraction, ventricular synchrony and sinus node dysfunction in the world.

So SJM China will sponsor a prospective, randomized, double blinded, multi-center, controlled study to evaluate the clinical impact at 18 months after DDD implantation of alternative pacing site (RVOTs and RVA) and the different conduction path (RVOTs and AV node) on cardiac dysfunction prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with only sinus-node dysfunction and meet pacing indication
* Patients with LVEF≥60% and with ventricular synchrony.
* Patients signed the written informed consent for the study
* Patients can endure the required follow up

Exclusion Criteria:

* Patients with atrial fibrillation
* Patients with atrial-ventricular block
* Patients with LBBB
* Patients with significant valvular disease
* Patients with severe hematopathy or severe renal inadequacy
* Patients with life expectancy < 1.5 year
* Patients who are in the period of pregnant or lactation
* Patients who are younger than 18 years old
* Patients who are ongoing other devices or agents study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 18 months
  To demonstrate:
  * Whether RVOTs pacing is superior to right ventricular apical pacing in preserving left ventricular systolic function in patients with a normal left ventricular ejection fraction, ventricular synchrony and standard indications for pacing(sinus node dysfunction)
  * Whether RVOTs pacing is not inferior to AAI pacing in preserving left ventricular systolic function in patients with a normal left ventricular ejection fraction, ventricular synchrony and sinus node dysfunction.

SECONDARY OUTCOMES:
left ventricular end-systolic volume (LVESV) | 18 months
  To demonstrate:
  * Whether RVOTs pacing is superior to right ventricular apical pacing in avoiding adverse left ventricular remodeling in patients with a normal left ventricular ejection fraction, ventricular synchrony and standard indications for pacing(sinus node dysfunction)
  * Whether RVOTs pacing is not inferior to AAI pacing in avoiding adverse left ventricular remodeling in patients with a normal left ventricular ejection fraction, ventricular synchrony and sinus node dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang Dong General Hospital, Guangzhou, Guangdong, China